CLINICAL TRIAL: NCT04821843
Title: Cohort Study of Neoadjuvant Treatment Modalities for Esophageal Cancer
Brief Title: Neoadjuvant Treatment Modalities in Esophageal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XIN WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2721
Record Dates: First submitted 2021-03-15; First posted 2021-03-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Cancer; Chemotherapy Effect; Chemoradiation; Surgery; Targeted Therapy; Immunotherapy; Esophagogastric Juction Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Platinum Compounds; Surgical Procedures, Operative; Immunotherapy; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Neoadjuvant chemotherapy) nCT (Experimental): This arm received chemotherapy with or without immunotherapy/targeting agents as neoadjuvant treatment.
  Interventions: Drug: Platinum based chemotherapy; Drug: Paclitaxel based chemotherapy; Radiation: Radiotherpay; Procedure: Surgery; Drug: Immunotherapy; Drug: 5-FU Analog based chemotherpay; Drug: Nimotuzumab
- (Neoadjuvant Chemoradiation) nCRT (Placebo Comparator): This arm received chemoradiotherapy with or without immunotherapy/targeting agents as neoadjuvant treatment.
  Interventions: Drug: Platinum based chemotherapy; Drug: Paclitaxel based chemotherapy; Procedure: Surgery; Drug: Immunotherapy; Drug: 5-FU Analog based chemotherpay; Drug: Nimotuzumab

INTERVENTIONS:
Drug: Platinum based chemotherapy — q1-3W according to physician's preference
Drug: Paclitaxel based chemotherapy — q1-3W according to physician's preference
Radiation: Radiotherpay — 40-50Gy/1.8-2.2Gy/20-25f
  Arms: (Neoadjuvant chemotherapy) nCT
Procedure: Surgery — Radical esophagectomy
Drug: Immunotherapy — Anti-PD-1/PD-L1 Antibody
Drug: 5-FU Analog based chemotherpay — W1-5 qW or d1-14, q3W according to physician's preference
Drug: Nimotuzumab — 200-400mg, d1,qW

SUMMARY:
Esophageal cancer is the most prevalent cancer globally with poor survival outcome. The prognosis with surgery alone is poor, accounting for 30-40% of overall survival at 5 year. Either neoadjuvant chemotherapy (nCT) or chemoradiotherapy (nCRT) has been shown as efficatious therapy to improve patients outcomes in esophageal or esophagogastric junction cancer as compared with surgery alone. The purpose of this study was to explore the optimal neoadjuvant treatment modalities including PD-1/PD-L1 antibody or targeted drug for patients with esophageal or esophagogastric junction cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years；
* Esophageal or Esophagogastric cancer；
* Histologically proven squamous cell carcinoma or adenocarcinoma in patients staged as I-IVa (AJCC 8th)；
* Primary treatment performed in Cancer Hospital, Chinese Academy of Medical Sciences；
* ECOG PS score: 0~1；
* Estimated survival time ≥3 months；
* Normal organ and marrow function as defined below:Hemoglobin: greater than or equal to 100g/L ;Leukocytes: greater than or equal to 4,000 G/L; Neutrophil: greater than or equal to 2,000 G/L; Platelets: greater than or equal to 100,000/mm3 ; Creatinine: less than or equal to 1.5 times the upper limit or CCR greater than or equal to 60 ml/min; AST/ALT: less than or equal to 2.5 times the upper limit; Total bilirubin: less than or equal to 1.5 times the upper limit; INR: less than or equal to 1.5 times the upper limit; APTT: less than or equal to 1.5 times the upper limit; PT: less than or equal to 1.5 times the upper limit；
* Informed consent；

Exclusion Criteria:

* With any distant metastasis out of regional lymphatic drainage or in liver, lung, bone, CNS, etc；
* Patients with other cancer history in 5 years except cervical carcinoma in situ and non-malignant melanoma skin cancer；
* Existing active infection such as active tuberculosis and hepatitis；
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia；
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness History of allergic reactions attributed to paclitaxel, albumin or cisplatin；
* Participation in other clinical trials currently or within 4 weeks of selection；
* Pregnant or lactating females；
* Absence of medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2002-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 year

SECONDARY OUTCOMES:
Progression free survival | 1 year, 2 year, 3 year, 5 year
Number of participants with Acute and late toxicities of radiotherapy,chemotherapy and immunotherapy | 3 months
  Acute and late toxicities are evaluated by NCI-CTC version 5.0
Pathological response rate | 3 months
  Pathological response were classiﬁed into three grades.Grade I signiﬁes that there is little shrinkage in the tumor; only mild regression in the tumor cells is observed under themicroscope. Grade II shows gross reduction in size of the tumor and marked regression in the cancer cells microscopically, yet viable nests of cancer tissue are still visible. Grade III implies complete or almost total resolution of the tumor on exploration, and disappearance of the tumor tissue microscopically; only remnants of degenerated cancer cells can be seen (so-called ghost cancer cells).
R0 resection rate | 3 months
Locoregional recurrence free survival | 1 year, 2 year, 3 year, 5 year
Distant metastasis free survival | 1 year, 2 year, 3 year, 5 year

OTHER OUTCOMES:
Analysis of the correlation between radiation dose and the number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 1 year, 2 year, 3 year, 5 year
Radiomics analysis | 1 year, 2 year, 3 year, 5 year
  The value of Radiomics of MRI and CT in predicting pathological complete response (pCR) or no response (NR) and the correlation between radiomics of MRI and CT and overall survival (OS), which is defined as the time from the beginning of neoadjuvant chemotherapy to the death with any causes.
Target dealineation of organs at risk and their impact on the prognosis and adverse effects of radiotherapy | 1 year, 2 year, 3 year, 5 year
Target dealineation of clinical target volumn and their impact on the prognosis | 1 year, 2 year, 3 year, 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China